CLINICAL TRIAL: NCT05107310
Title: SpiNav - SPInal NAVigation Trial
Brief Title: The Spinal Navigation Trial - Surgical Navigation or Free Hand Technique in Spine Surgery
Acronym: SPINAV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Uppsala University (Other)
Responsible Party: Principal Investigator, Paul Gerdhem, Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPINAV
Record Dates: First submitted 2021-09-14; First posted 2021-11-04 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Scoliosis; Kyphosis
MeSH Terms: conditions — Scoliosis; Kyphosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Navigation group 1 ARSN (Experimental): Augmented reality surgical navigation (ARSN). Pedicle screw placement using the Philips ClarifEye system combined with Philips Allura for imaging.
  Interventions: Procedure: Pedicle screws insertion using ARSN
- Control group 1 FH (Active Comparator): Free hand (FH) surgical technique. Pedicle screw placement using conventional free hand technique.
  Interventions: Procedure: Pedicle screws insertion by free hand technique
- Navigation group 2 IRSN (Experimental): Infrared surgical navigation (IRSN). Pedicle screw placement using Brainlab Curve 1.2 combined with Medtronic o-arm for imaging.
  Interventions: Procedure: Pedicle screws insertion using IRSN
- Control group 2 FH (Active Comparator): Free hand (FH) surgical technique. Pedicle screw placement using conventional free hand technique.
  Interventions: Procedure: Pedicle screws insertion by free hand technique

INTERVENTIONS:
Procedure: Pedicle screws insertion by free hand technique — Spinal deformity correction. Pedicle screws are inserted using free hand technique with the help of intraoperative fluoroscopy if needed.
  Arms: Control group 1 FH; Control group 2 FH
Procedure: Pedicle screws insertion using ARSN — Spinal deformity correction. Pedicle screws are inserted using augmented reality surgical navigation (ARSN) with the ClarifEye navigation system and the Philips Allura 2D/3D imaging system.
  Arms: Navigation group 1 ARSN
Procedure: Pedicle screws insertion using IRSN — Spinal deformity correction. Pedicle screws are inserted using infra-red surgical navigation (IRSN) with the Brainlab Curve 1.2 navigation system combined with the Medtronic O-arm 2D/3D imaging system.
  Arms: Navigation group 2 IRSN

SUMMARY:
The spinal navigation trial (SPINAV) is a randomized controlled trial (RCT) evaluating the use of computer-assisted navigation in surgery for spinal deformity

DETAILED DESCRIPTION:
Spinal deformity is a common reason for spinal surgery at youth. In addition, the incidence of surgery for spinal deformity in older adults is increasing. Spinal deformity surgery is by far the most complex spine surgery. One complexity lies in the correct placement of implants in the severely deformed spine. Today, the most common surgical procedures for spinal deformity involve placement of screws in the vertebral pedicle in the instrumented part of the spine. This gives good bone purchase, which is important for deformity correction.

The pedicle is narrow and misplaced pedicle screws can result in vascular, pulmonary or neural injuries, or inadequate bone purchase. Compared to the conventional free-hand surgical technique, which relies on the knowledge of anatomy, computer-assisted navigation using intraoperative 3D imaging has been shown to improve screw placement accuracy and reduce complications due to screw misplacements. As a consequence, navigation may also reduce the frequency of postoperative revision surgery compared to free hand. However, navigation still takes time, and is associated with higher intraoperative radiation than the free hand technique.

As of yet, the majority of data in this area are based on retrospectively collected series, and some prospectively collected series, while randomized controlled trials on spinal deformity are lacking.

In this randomized controlled trial the accuracy of pedicle screw placement using augmented reality surgical navigation (ARSN), infra-red surgical navigation (IRSN) and conventional free-hand technique will be investigated.

Patients of age 12 years and older with spinal deformities are randomized into one of the three surgical techniques mentioned above.

The primary outcome variable is pedicle screw placement accuracy at 1st attempt assessed using the Gertzbein scale.

Data from the navigated groups (ASRN and IRSN) will be analyzed together, and compared with the free hand groups analyzed together. The ASRN and ISRN groups will also be compared with their respective free hand groups.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by patient or legal guardian
* Age 12 years and older
* Spinal deformity surgery

Exclusion Criteria:

* Unable to give informed consent
* Surgery without pedicle screws
* Previous surgery with pedicle screws in the planned surgical area

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Accurately placed pedicle screws | Intraoperative
  The primary endpoint is the percentage of accurately placed pedicle screws assessed using the Gertzbein scale and based on intraoperative verification scan cone beam computed tomography (CBCT).

SECONDARY OUTCOMES:
Pedicle screw intraoperative revision rates-clinical assessment | Intraoperative
  Number of screws intraoperatively revised based on clinical assessment
Pedicle screw intraoperative revision rates- neurophysiology | Intraoperative
  Number of screws intraoperatively revised based on neurophysiology
Pedicle screw intraoperative revision rates- intraoperative verification | Intraoperative
  Number of screws intraoperatively revised based on intraoperative verification CBCT scan
Accuracy for ARSN - path deviation in mm | Intraoperative
  Deviation from planned navigated path in mm at bone entry and screw tip measured on the postoperative computed tomography (CT)
Accuracy for IRSN- path deviation in mm | Intraoperative
  Deviation from navigated path in mm at bone entry and screw tip measured on the postoperative computed tomography (CT)
Accuracy for ARSN - angular deviation | Intraoperative
  Angular deviation (degrees) of the placed screw compared to the planned navigated path measured on the postoperative computed tomography (CT)
Accuracy for IRSN - angular deviation | Intraoperative
  Angular deviation of the placed screw compared to the navigated path measured on the postoperative computed tomography (CT)
Accuracy at 1st attempt | Intraoperative
  Accuracy at 1st attempt = (Screws placed at first attempt according to intraoperative protocols and graded 0 or 1) / (total number of placed screws).
  Assessed on intraoperative CBCT
Final accuracy of placed pedicle screws | Intraoperative
  Final accuracy of placed pedicle screws is calculated as: number of accurately placed screws (Gertzbein grade 0+1) according to postoperative CT / total number of placed screws.
Pedicle screw placement density | Intraoperative
  The study aims for 100% pedicle screw density. Hooks may be placed as rescue or if screw placement fails.
Pedicle screw placement in relation to morphometric measurements | Preoperative and intraoperative
  Pedicle diameters are measured on preoperative and intraoperative CT. Pedicle screw placement measured on intraoperative and postoperative CT.
Deformity correction change | 3-6 months post-op
  Cobb angle change from preoperative to first erect postoperative radiograph
Patient radiation dose exposure | Intraoperative
  Patient radiation exposure (ED in mSv) for the whole procedure, Patient radiation exposure (ED in mSv) for fluoroscopy Patient radiation exposure (ED in mSv) for each CBCT
Staff radiation dose exposure | Intraoperative
  Average staff radiation exposure (in mSv) for the whole procedure
Intraoperative characteristics- procedure time | Intraoperative
  Total procedure time as well as normalized to number of spinal levels from the upper to the lower instrumented vertebra.
Intraoperative characteristics- planning time | Intraoperative
  Intraoperative planning time (from start of planning in navigation software until last screw planned) (only when treated with ARSN or IRSN)
Intraoperative characteristics- instrumentation time | Intraoperative
  Instrumentation time (total time for navigated/FH screw placement from first to last screw placement)
Intraoperative characteristics- instrumentation time/level | Intraoperative
  Instrumentation time normalized to number of levels
Intraoperative characteristics- time for verification imaging | Intraoperative
  Time for intraoperative verification imaging (CBCT and/or Fluoroscopy)
Intraoperative characteristics- screw placement time | Intraoperative
  Screw placement time (per screw, from start with awl to screw placed)
Intraoperative characteristics- blood loss | Intraoperative
  Intraoperative blood loss
Inpatient stay | Measured from day of surgery until day of discharge. Usual length of stay is less than one week, and maximum two weeks.
  Length of hospital stay in days
Patient reported outcome measures- Scoliosis Research Society 22 revised (SRS-22r) | up to 5 years
  The scoliosis specific questionnaire SRS-22r ranging from 1 (worst) to 5 (best)
Patient reported outcome measures- the 24 item Early Onset Scoliosis Questionnaire (EOSQ-24) | up to 5 years
  The scoliosis specific questionnaire EOSQ-24 ranging from 0 (worst) to 100 (best)
Patient reported outcome measures- Oswestry Disability Index (ODI) | up to 5 years
  The back disabiliy questionnaire (ODI) ranging from 0 (best) to 100 (worst)
Patient reported outcome measures- EQ-5D 3 level version (EQ-5D-3L) | up to 5 years
  The generic quality of life EQ-5D-3L index ranging from -0.59 (worst) to 1.00 (best)
Complications | At 30 days, at 90 days
  Number of patients that have had complications
Revision surgery | At 30 days, at 90 days, at 1 year
  Number of patients that have undergone revision surgeries
Cost per patient | At 30 days, at 90 days, at 1 year
  Cost per patient

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gerdhem, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Manuscripts will be submitted for publication in peer-reviewed journals. Quality-controlled raw data as well as processed data used in publications will be made available at the time of publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The detailed protocol, including the statistical analysis plan will be submitted for publication after study start. No end date.
Access Criteria: Either as an appendix to publications, or at a repository at the Sponsor of the trial.

REFERENCES:
- [Derived] El-Hajj VG, Charalampidis A, Fell D, Edstrom E, Elmi-Terander A, Gerdhem P. Study protocol: the SPInal NAVigation (SPINAV) trial - comparison of augmented reality surgical navigation, conventional image-guided navigation, and free-hand technique for pedicle screw placement in spinal deformity surgery. BMC Musculoskelet Disord. 2025 Jun 2;26(1):543. doi: 10.1186/s12891-025-08817-3. PMID 40457280